CLINICAL TRIAL: NCT03844919
Title: TICS: Transcranial Magnetic Stimulation for Intervening in Children With Tourette's Syndrome
Brief Title: TICS: Transcranial Magnetic Stimulation for Intervening in Children With Tourette's Syndrome (CIHR)
Acronym: TICS-CIHR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Frank MacMaster, PhD, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB18-0220
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Tic Disorders
Keywords: Children; Adolescent; CBIT; Transcranial magnetic stimulation; Comprehensive Behavioral Intervention for Tics; rTMS; TMS; MRI; Tourette's Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Children (N = 50, 6-18 years) with TS will be randomized to either a (1) rTMS+CBIT arm, or a (2) sham rTMS+CBIT arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible subjects will be randomly assigned to receive one of the two treatment regimens in a 1:1 ratio. Dr. Nettel-Aguirre will generate the sequence with random sized blocks of 2,4 and 6 and use the REDCap randomization module for recruiters to access the allocation for the subjects. The algorithm will stratify each by sex and age group (6-10, 11-14, 15-18 years). Dr. Zewdie will set up the rTMS accordingly for active or sham delivery. Participants and their parents will be blind to group status regarding sham vs. active rTMS. Dr. Wilcox, and all raters responsible for clinical evaluation under Dr. Wilcox's supervision, will also be blinded to group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS + CBIT (Experimental): Repetitive transcranial magnetic stimulation (rTMS) and Comprehensive Behavioural Intervention for Tics (CBIT)
  Interventions: Device: rTMS + CBIT; Behavioral: Sham rTMS + CBIT
- Sham rTMS + CBIT (Active Comparator): Sham repetitive transcranial magnetic stimulation (rTMS) and Comprehensive Behavioural Intervention for Tics (CBIT)
  Interventions: Behavioral: Sham rTMS + CBIT

INTERVENTIONS:
Device: rTMS + CBIT — Repetitive Transcranial Magnetic Stimulation (rTMS) parameters are: intensity 100% resting motor threshold (RMT), frequency 1Hz, duration = 30 minutes (1800 stimulations; 900 per side), target - the supplementary motor area (SMA). Treatments occur on weekdays (T - F) for four weeks (20 total).
  The Comprehensive Behavioral Intervention for Tics (CBIT) will be completed over eight sessions that will average 60 minutes in duration. First, participants will undergo awareness training. Participants will then be introduced to competing response training, which involves performing a voluntary behaviour designed to disrupt the execution of the tic. The eight sessions will occur on Mondays, once a week for six weeks and then on weeks 8 and 10.
  Arms: rTMS + CBIT
Behavioral: Sham rTMS + CBIT — Sham rTMS (sham coil) will be paired with CBIT. Sham rTMS will be delivered over the same time-frame as above. CBIT will be identical to the above.

SUMMARY:
Tourette's Syndrome (TS) is characterized by repetitive movements and vocalizations called tics. Due to the suffering caused by TS, children and adolescents often require treatment for their tics. The investigators' research focuses on developing novel repetitive transcranial magnetic stimulation (rTMS) interventions for child and adolescent neuropsychiatric disorders. In this project, the investigators will determine the effect of pairing 3 weeks of rTMS and HRT on tic severity and plasticity as indexed by supplementary motor area (SMA) y-aminobutyric acid (GABA) concentration and functional connectivity of the SMA to the primary motor cortex (M1) in children and adolescents with TS.

Children (N = 50, 6-18 years) with TS will be randomized to either a (1) rTMS+HRT arm, or (2) sham rTMS+HRT. Outcome measures will examine tic severity (primary), brain chemistry and function (secondary) at baseline and then at week 7. The investigators' proposed aims are:

(Aim 1) To determine the effect of paired rTMS and HRT on tic severity as measured by the Yale Global Tic Severity Scale (YGTSS) by comparing it to sham rTMS + HRT.

1-1: The investigators hypothesize that tic severity will decrease from baseline to post-treatment.

1-2: The investigators also hypothesize that the reduction in tic severity will be greater in the paired treatment group (rTMS+HRT > Sham rTMS+HRT).

(Aim 2) To determine the effect of paired rTMS and HRT on brain plasticity compared to sham rTMS + HRT.

2-1: The investigators hypothesize that patients treated with the paired rTMS and HRT will have a greater increase in GABA concentration comparted to sham and HRT.

2-2: The investigators also hypothesize that functional connectivity between the SMA and M1 will be greater with paired treatment (rTMS+HRT > Sham rTMS+HRT).

DETAILED DESCRIPTION:
Tourette's Syndrome (TS) is characterized by repetitive movements and vocalizations called tics. Due to the suffering caused by TS, children and adolescents often require treatment for their tics. Tic severity predicts poor outcomes across physical, psychological, and cognitive domains in youth. Current treatments for TS remain limited in scope and efficacy. Atypical antipsychotics are often used and for many patients have an unacceptable side effect burden. Behavioral treatments, like habit reversal therapy (HRT), show promise and are safe, but are predicated on a certain level of brain maturation to execute.

The investigators' research focuses on developing novel repetitive transcranial magnetic stimulation (rTMS) interventions for child and adolescent neuropsychiatric disorders. Plasticity, precision, and pairing are key considerations in this process. In this project, the investigators will determine the effect of pairing 3 weeks of rTMS and HRT on tic severity and plasticity as indexed by supplementary motor area (SMA) y-aminobutyric acid (GABA) concentration and functional connectivity of the SMA to the primary motor cortex (M1) in children and adolescents with TS. The investigators will use functional magnetic resonance imaging (fMRI) and robot controlled rTMS to precisely target the SMA. The investigators believe this pairing will provide improved relief by inducing plasticity to retrain the brain to be better at suppressing tics at an earlier age than usually expected.

Children (N = 50, 6-18 years) with TS will be randomized to either a (1) rTMS+HRT arm, or (2) sham rTMS+HRT. Outcome measures will examine tic severity (primary), brain chemistry and function (secondary) at baseline and then at week 7. The investigators' proposed aims are:

(Aim 1) To determine the effect of paired rTMS and HRT on tic severity as measured by the Yale Global Tic Severity Scale (YGTSS) by comparing it to sham rTMS + HRT.

1-1: The investigators hypothesize that tic severity will decrease from baseline to post-treatment.

1-2: The investigators also hypothesize that the reduction in tic severity will be greater in the paired treatment group (rTMS+HRT > Sham rTMS+HRT).

(Aim 2) To determine the effect of paired rTMS and HRT on brain plasticity compared to sham rTMS + HRT.

2-1: The investigators hypothesize that patients treated with the paired rTMS and HRT will have a greater increase in GABA concentration comparted to sham and HRT.

2-2: The investigators also hypothesize that functional connectivity between the SMA and M1 will be greater with paired treatment (rTMS+HRT > Sham rTMS+HRT).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Tourette's syndrome
2. IQ greater than 80
3. English fluency (to enable assent and consent).

Exclusion Criteria:

1. Diagnosis of mania or schizophrenia
2. Impediments to TMS or MRI.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale Total Tic score (YGTSS) | Baseline to week 7
  30% reduction in Yale Global Tic Severity Scale Total Tic score (YGTSS) (~9 point reduction).
  A higher score on all scales suggests a more severe tics.
  The YGTSS provides two tic severity scores:
  1. Total Motor (0 to 25)
  2. Total Phonic (0 to 25)
  These are summed to form the Total Tic Severity Score (0 to 50). This is the measure for the primary outcome variable.
  There is also the separate Impairment Dimension Score (0 to 50).
  The total score is hence 0 to 100 (sum of Total Tic Severity Score and Impairment Dimension Score).

SECONDARY OUTCOMES:
Supplementary Motor Area (SMA) GABA concentration as measured by LCModel (Institutional Units) | Baseline to week 7
  10% increase in GABA concentration in the Supplementary Motor Area (SMA) as measured by LCModel (Institutional Units)
Functional connectivity of the Supplementary Motor Area (SMA) and the dominant Primary Motor Cortex (M1) | Baseline to week 7
  Functional connectivity, as measured using SPM12, of the Supplementary Motor Area (SMA) and the dominant Primary Motor Cortex (M1).

OTHER OUTCOMES:
Yale Global Tic Severity Scale Total Tic score (YGTSS) post CBIT | Baseline to week 11
  30% reduction in YGTSS (~9 point reduction)
  30% reduction in Yale Global Tic Severity Scale Total Tic score (YGTSS) (~9 point reduction).
  A higher score on all scales suggests a more severe tics.
  The YGTSS provides two tic severity scores:
  1. Total Motor (0 to 25)
  2. Total Phonic (0 to 25)
  These are summed to form the Total Tic Severity Score (0 to 50). This is the measure for this outcome variable.
  There is also the separate Impairment Dimension Score (0 to 50).
  The total score is hence 0 to 100 (sum of Total Tic Severity Score and Impairment Dimension Score).

CONTACTS AND LOCATIONS:
Overall Officials: Frank P MacMaster, PhD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data would be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, and ICF is open to be shared now. De-identified data will be shared after we submitted our main papers. This is estimated in 2025.
Access Criteria: Email for permission from PI of project.

REFERENCES:
- [Derived] Kahl CK, Swansburg R, Kirton A, Pringsheim T, Wilcox G, Zewdie E, Harris A, Croarkin PE, Nettel-Aguirre A, Chenji S, MacMaster FP. Targeted Interventions in Tourette's using Advanced Neuroimaging and Stimulation (TITANS): study protocol for a double-blind, randomised controlled trial of transcranial magnetic stimulation (TMS) to the supplementary motor area in children with Tourette's syndrome. BMJ Open. 2021 Dec 24;11(12):e053156. doi: 10.1136/bmjopen-2021-053156. PMID 34952879